CLINICAL TRIAL: NCT04760262
Title: The Effect of Different Anesthesia Techniques on Cerebral Oxygenation in Thoracic Surgery
Brief Title: The Effect of Anesthesia on Cerebral Oxygenation
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Ali AKDOĞAN, assistant professor, Karadeniz Technical University
Other Study IDs: 2013/21
Record Dates: First submitted 2021-02-10; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: One-Lung Ventilation; Thoracic Surgery; Postoperative Cognitive Complications
Keywords: One-lung ventilation; cerebral oxygenation; postoperative cognitive dysfunction; sevoflurane; propofol
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Sevoflurane; Propofol; Remifentanil

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group Propofol: anesthesia was maintained with TIVA (intravenous 125-250 µg/kg/min propofol + 0.1-0.25 µg/kg/min remifentanil infusion)
  Interventions: Drug: Propofol
- Group Sevoflurane: anesthesia was maintained with inhalation (sevoflurane concentration of 1-2% in 50-50% O2-air mixture).
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane %2-3 for general anesthesia maintenance, BIS values were arranged 40-60 until the end of operation, In case of tachycardia or hypertension the opioid dose was reduced, in case of bradycardia or hypertension the opioid dose was increased
  Groups: Group Sevoflurane
Drug: Propofol — BIS values were arranged 40-60 until the end of operation, In case of tachycardia or hypertension the opioid dose was reduced, in case of bradycardia or hypertension the opioid dose was increased
  Other Names: Remifentanil
  Groups: Group Propofol

SUMMARY:
One-lung ventilation (OLV) may cause negative changes in the oxygenation of cerebral tissue which results in postoperative cognitive dysfunction. The aim of this prospective study was to compare the potential effects of TIVA and inhalation general anesthesia techniques on cerebral tissue oxygenation and postoperative cognitive functions in patients receiving one-lung ventilation in thoracic surgery

DETAILED DESCRIPTION:
One-lung ventilation (OLV) is a commonly used technique in thoracic surgeries. In thoracic surgeries performed with OLV, there may be changes in cerebral tissue oxygenation depending on both patient position and anesthetic technique. The effect of cerebral hypoxia on postoperative cognitive functions is controversially. Despite the ISPOCD1 study in which concluded that there were no relationship between the cerebral hypoxy and postoperative cognitive dysfunction (POCD) regional cerebral oxygen saturation decrements during surgery are listed among the POCD When OLV begins, alveolar hypoxia and arteriovenous shunt of deoxygenated blood occur in the dependant lung. And then, hypoxic pulmonary vasoconstriction (HPV) in non-ventilated lung segments occurs with increased mechanical stress. This event lead to significant physiological changes in cardiac output and pulmonary and systemic pressures In OLV, the propofol-based total intravenous anesthesia (TIVA) and inhalation general anesthesia techniques are frequently used. Recent studies have shown that unlike inhalational anesthetics, propofol does not suppress HPV, indeed increases it (Inhalational anesthetic agents reduce cardiac output more than oxygen consumption, causing a decrease in mixed venous partial pressure of oxygen, which stimulates hypoxic pulmonary vasoconstriction . Studies have shown significant reductions in cerebral oxygen saturation in thoracic surgery as a result of severe oxidative stress due to prolonged OLV and hypoxemia due to decreased functional residual capacity of the ventilated lung in the lateral decubitus position Cerebral oximetry is a method used to monitor the cerebral oxygen distribution-consumption balance and regional oxygen saturation (rSO2) in a limited area of the frontal cortex by noninvasively and continuously combining arterial and venous oxygen saturation signals of near-infrared spectroscopy (NIRS), which is a technique developed in the 1970s. Thanks to this method, perioperative physiological conditions, optimal tissue oxygenation and end-organ functions can be interpreted The aim of this prospective study was to compare the potential effects of TIVA and inhalation general anesthesia techniques on cerebral tissue oxygenation and postoperative cognitive functions in patients receiving one-lung ventilation in thoracic surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients in American Society of Anesthesiology (ASA) classification I and II
* Patients who would undergo thoracic surgery with one-lung ventilation (OLV)
* thoracic surgeries with one-lung ventilation (OLV) that will take at least 45 minutes

Exclusion Criteria:

* Patients in ASA classification III and higher
* Emergency surgery
* Patients with known allergy to drugs used in the study
* Patients in New York Heart Association classification III-IV
* severe metabolic, renal, hepatic, central nervous system diseases, alcohol or drug addiction
* multiple trauma, coagulapathy, cerebral disease, dementia, hearing impairment and imperception
* severe obesity (a body mass index (BMI) of ≥ 35)
* patients with a peripheral oxygen saturation below 90 during one lung ventilation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who would undergo thoracic surgery with one-lung ventilation (OLV)
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Near Infrared Spectroscopy | Duration of surgery
  Cerebral oxygen saturation as measured by Near Infrared Spectroscopy
Mini mental state examination (MMSE) | 3 to 24 hours postoperative period
  Mini mental state examination (MMSE) to evaluate patients' cognitive functions

SECONDARY OUTCOMES:
mean arterial pressure | Duration of surgery
  The effect of anesthetics on mean arterial pressure
heart rate | Duration of surgery
  The effect of anesthetics on heart rate
bispectral index | Duration of surgery
  The effects of sevoflurane and desflurane on bispectral index

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

REFERENCES:
- [Background] Hood R, Budd A, Sorond FA, Hogue CW. Peri-operative neurological complications. Anaesthesia. 2018 Jan;73 Suppl 1:67-75. doi: 10.1111/anae.14142. PMID 29313909
- [Background] Nakayama M, Murray PA. Ketamine preserves and propofol potentiates hypoxic pulmonary vasoconstriction compared with the conscious state in chronically instrumented dogs. Anesthesiology. 1999 Sep;91(3):760-71. doi: 10.1097/00000542-199909000-00029. PMID 10485788
- [Background] Kazan R, Bracco D, Hemmerling TM. Reduced cerebral oxygen saturation measured by absolute cerebral oximetry during thoracic surgery correlates with postoperative complications. Br J Anaesth. 2009 Dec;103(6):811-6. doi: 10.1093/bja/aep309. PMID 19918024
- [Background] Mahal I, Davie SN, Grocott HP. Cerebral oximetry and thoracic surgery. Curr Opin Anaesthesiol. 2014 Feb;27(1):21-7. doi: 10.1097/ACO.0000000000000027. PMID 24263686
- [Background] Aguirre JA, Marzendorfer O, Brada M, Saporito A, Borgeat A, Buhler P. Cerebral oxygenation in the beach chair position for shoulder surgery in regional anesthesia: impact on cerebral blood flow and neurobehavioral outcome. J Clin Anesth. 2016 Dec;35:456-464. doi: 10.1016/j.jclinane.2016.08.035. Epub 2016 Oct 18. PMID 27871574